CLINICAL TRIAL: NCT01703286
Title: Randomized, Three Period Cross Over, Double Blind, Double Dummy Study in Type 2 Diabetic Patients to Assess the Endothelial Effects of Linagliptin, Glimepiride and Placebo Therapy for 28 Days ('ENDOTHELINA')
Brief Title: Trial to Assess the Influence of 4 Weeks' Treatment With Linagliptin as Compared to Glimepiride and Placebo on Endothelial Function in Patients With Type 2 Diabetes Using FMD (Flow-Mediated Vasodilation)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.105; 2012-003317-33 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-10-01; First posted 2012-10-10 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin; glimepiride

ARMS (3):
- Linagliptin 5mg (Experimental): given once daily over 28 days
  Interventions: Drug: Placebo; Drug: Linagliptin
- Glimepiride (Active Comparator): given once daily in 1mg dosis over 7 days, following a titration step to 2mg and application for 21 days
  Interventions: Drug: Placebo; Drug: Glimepiride
- Placebo (Placebo Comparator): given once daily over 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo matching Glimepiride
  Arms: Linagliptin 5mg
Drug: Linagliptin — given once daily for 28 days
  Arms: Linagliptin 5mg
Drug: Placebo — Placebo matching Linagliptin
  Arms: Glimepiride
Drug: Placebo — Placebo matching Linagliptin
  Arms: Placebo
Drug: Placebo — Placebo matching Glimepiride
  Arms: Placebo
Drug: Glimepiride — 1 mg for 7 days followed by uptitration to 2 mg (given for following 21 days)
  Arms: Glimepiride

SUMMARY:
The general aim of the present study is to investigate the impact of 4 weeks treatment with linagliptin (5 mg) on endothelial function in patients with type 2 diabetes mellitus. In the current trial this effect of linagliptin treatment on endothelial function will be compared against both the sulfonylurea glimepiride and against placebo, which has not been tested in a trial before; as also is the case for other DPP-4 inhibitors.

Besides placebo, glimepiride was chosen as a comparator, as it is one compound of the second most used oral antidiabetic drug class.

ELIGIBILITY:
Inclusion criteria:

1. Type 2 diabetic male and female patients according to the following criteria:

   Based upon a complete medical history and clinical laboratory tests
2. Age >= 18 and Age <= 65 years
3. Body mass index >= 25 <= 35 kg/m2
4. HbA1c <= 7.5%
5. Treatment with metformin (=1500 mg daily) for <= 3 months
6. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation.

   For female patients of childbearing potential:
7. Use of acceptable method of contraception (Pearl-Index <1).

Exclusion criteria:

1. Treatment with any glucose-lowering drug except for metformin within prior 3 months.
2. Any finding of the medical examination (including blood pressure, pulse rate and electrocardiogram) deviating from normal and of clinical relevance.
3. Any evidence of a clinically relevant acute concomitant disease
4. History of cardiovascular disease (e.g. coronary artery disease history of acute myocard infarction or stroke, peripheral vascular disease).
5. History of major diabetic complications (e.g. nephropathy, retinopathy)
6. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, immunological or hormonal disorders (except: hypertension treated with angiotensin receptor blocker or angiotensin-converting-enzyme inhibitors, hyperlipidemia with statin therapy, thyroid hormone replacement therapy, all stable for at least three months prior to screening).
7. Surgery of the gastrointestinal tract (except appendectomy).
8. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders.
9. History of relevant orthostatic hypotension, fainting spells or blackouts.
10. Chronic or relevant acute infections.
11. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients).
12. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial.
13. Participation in another trial with an investigational drug within one month prior to administration or during the trial.
14. Smoker (>= 1 cigarettes or >= 1 cigars or >= 1 pipes/day).
15. Alcohol abuse (more than 60 g/day).
16. Drug abuse.
17. Blood donation (more than 100 mL within four weeks prior to administration or during the trial).
18. Excessive physical activities (within one week prior to administration or during the trial).
19. Any laboratory value outside the reference range that is of clinical relevance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1218.105.001 Boehringer Ingelheim Investigational Site, Neuss, Germany

REFERENCES:
- [Derived] Jax T, Stirban A, Terjung A, Esmaeili H, Berk A, Thiemann S, Chilton R, von Eynatten M, Marx N. A randomised, active- and placebo-controlled, three-period crossover trial to investigate short-term effects of the dipeptidyl peptidase-4 inhibitor linagliptin on macro- and microvascular endothelial function in type 2 diabetes. Cardiovasc Diabetol. 2017 Jan 21;16(1):13. doi: 10.1186/s12933-016-0493-3. PMID 28109295

RESULTS

PARTICIPANT FLOW:
Groups:
- Pbo/ G1-4/ L 5: Placebo tablet once daily over 28 days/ Glimepiride 1 tablet (1 mg) once daily for 7 days followed by uptitration to 2 to 4 mg once daily within next 21 days/ Linagliptin 1 tablet (5 mg) once daily for 28 days
- L 5/ G 1-4/ Pbo: Linagliptin 1 tablet (5 mg) once daily for 28 days/ Glimepiride 1 tablet (1 mg) once daily for 7 days followed by uptitration to 2 to 4 mg once daily within next 21 days/ Placebo tablet once daily over 28 days
- G 1-4/ L 5/ Pbo: Glimepiride 1 tablet (1 mg) once daily for 7 days followed by uptitration to 2 to 4 mg once daily within next 21 days/ Linagliptin 1 tablet (5 mg) once daily for 28 days/ Placebo tablet once daily over 28 days
- G1-4/ Pbo/ L 5: Glimepiride 1 tablet (1 mg) once daily for 7 days followed by uptitration to 2 to 4 mg once daily within next 21 days/ Placebo tablet once daily over 28 days/ Linagliptin 1 tablet (5 mg) once daily for 28 days
- Pbo/ L 5/ G1-4: Placebo tablet once daily over 28 days/ Linagliptin 1 tablet (5 mg) once daily for 28 days/ Glimepiride 1 tablet (1 mg) once daily for 7 days followed by uptitration to 2 to 4 mg once daily within next 21 days
- L 5/ Pbo/ G1-4/: Linagliptin 1 tablet (5 mg) once daily for 28 days/ Placebo tablet once daily over 28 days/ Glimepiride 1 tablet (1 mg) once daily for 7 days followed by uptitration to 2 to 4 mg once daily within next 21 days
Period: Period 1 Including Washout
Arm/Group | Pbo/ G1-4/ L 5 | L 5/ G 1-4/ Pbo | G 1-4/ L 5/ Pbo | G1-4/ Pbo/ L 5 | Pbo/ L 5/ G1-4 | L 5/ Pbo/ G1-4/
Started | 7 | 7 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1
Period: Period 2 Including Washout
Arm/Group | Pbo/ G1-4/ L 5 | L 5/ G 1-4/ Pbo | G 1-4/ L 5/ Pbo | G1-4/ Pbo/ L 5 | Pbo/ L 5/ G1-4 | L 5/ Pbo/ G1-4/
Started | 7 | 7 | 7 | 6 | 7 | 6
Completed | 7 | 7 | 7 | 5 | 7 | 6
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Period: Period 3 Including Washout
Arm/Group | Pbo/ G1-4/ L 5 | L 5/ G 1-4/ Pbo | G 1-4/ L 5/ Pbo | G1-4/ Pbo/ L 5 | Pbo/ L 5/ G1-4 | L 5/ Pbo/ G1-4/
Started | 7 | 7 | 7 | 5 | 7 | 6
Completed | 7 | 7 | 7 | 5 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: TS (treated set) - included all patients who were dispensed trial medication and were documented to have taken at least 1 dose of trial drug.
Groups:
- Total Participants: All study participants
Arm/Group | Total Participants
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Flow Mediated Vasodilation (FMD) Under Fasted Condition on Day 28
Description: Endothelial function under fasted condition was measured with flow mediated vasodilation (FMD). The change from baseline was calculated as the value on Day 28 divided by the respective value at baseline.
Time Frame: baseline and day 28 for each treatment arm
Population: Efficacy set (ES)- included all patients of the TS who provided at least 1 observation for at least 1 primary, secondary, or other efficacy endpoint without important protocol violations relevant for the statistical evaluation of these endpoints.
Measure: Geometric Mean (90% Confidence Interval); unit: percentage
Groups:
- Linagliptin 5 mg: Linagliptin: 1 tablet (5 mg) once daily for 28 days
- Glimepiride 1-4 mg: Glimepiride: 1 tablet (1 mg) once daily for 7 days followed by uptitration to 2 to 4 mg once daily within next 21 days
- Placebo: Placebo: matching Linagliptin or Glimepiride tablet once daily over 28 days
Arm/Group | Linagliptin 5 mg | Glimepiride 1-4 mg | Placebo
Number analyzed (Participants) | 39 | 41 | 39
percentage | 0.885 [0.695 to 1.128] | 1.002 [0.795 to 1.262] | 1.002 [0.786 to 1.277]
Statistical Analysis 1: Comparison: Linagliptin 5 mg vs Glimepiride 1-4 mg; Test type: Superiority or Other; p = 0.5403, ANOVA; Geometric mean ratio (net) = 0.884, 90% CI 2-sided [0.633 to 1.235]
Statistical Analysis 2: Comparison: Linagliptin 5 mg vs Placebo; Test type: Superiority or Other; p = 0.5402, ANOVA; Geometric mean ratio (net) = 0.884, 90% CI 2-sided [0.632 to 1.235]
Statistical Analysis 3: Comparison: Glimepiride 1-4 mg vs Placebo; Test type: Superiority or Other; p = 0.9989, ANOVA; Geometric mean ratio (net) = 1.000, 90% CI 2-sided [0.715 to 1.397]

2. Secondary Outcome: Change From Baseline in Flow Mediated Vasodilation (FMD) 2 h Post Meal on Day 28
Description: Endothelial function 2 hours post meal was measured with flow mediated vasodilation (FMD). The change from baseline was calculated as the value on Day 28 divided by the respective value at baseline.
Time Frame: baseline and day 28 for each treatment arm
Measure: Geometric Mean (90% Confidence Interval); unit: Percentage
Arm/Group | Linagliptin 5 mg | Glimepiride 1-4 mg | Placebo
Number analyzed (Participants) | 38 | 41 | 39
Percentage | 1.262 [0.968 to 1.646] | 1.045 [0.815 to 1.339] | 1.009 [0.777 to 1.311]
Statistical Analysis 1: Comparison: Linagliptin 5 mg vs Glimepiride 1-4 mg; Test type: Superiority or Other; p = 0.3885, ANOVA; Geometric mean ratio (net) = 1.208, 90% CI 2-sided [0.840 to 1.738]
Statistical Analysis 2: Comparison: Linagliptin 5 mg vs Placebo; Test type: Superiority or Other; p = 0.3105, ANOVA; Geometric mean ratio (net) = 1.251, 90% CI 2-sided [0.868 to 1.801]
Statistical Analysis 3: Comparison: Glimepiride 1-4 mg vs Placebo; Test type: Superiority or Other; p = 0.8749, ANOVA; Geometric mean ratio (net) = 1.035, 90% CI 2-sided [0.721 to 1.485]

3. Secondary Outcome: Change From Baseline in 2 Hours Post Meal Endothelial Independent Vasodilation (EIDV) on Day 28
Description: Endothelial function 2h post-meal was measured by endothelial independent vasodilation (EIDV). The change from baseline was calculated as the value on Day 28 divided by the respective value at baseline.
Time Frame: baseline and day 28 for each treatment arm
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: percentage
Arm/Group | Linagliptin 5 mg | Glimepiride 1-4 mg | Placebo
Number analyzed (Participants) | 39 | 41 | 39
percentage | 1.003 [0.945 to 1.061] | 1.053 [0.998 to 1.108] | 0.981 [0.923 to 1.039]
Statistical Analysis 1: Comparison: Linagliptin 5 mg vs Glimepiride 1-4 mg; Test type: Superiority or Other; p = 0.2982, ANOVA; Mean Difference (Net) = -0.050, 90% CI 2-sided [-0.130 to 0.030], Standard Error of Mean 0.048
Statistical Analysis 2: Comparison: Linagliptin 5 mg vs Placebo; Test type: Superiority or Other; p = 0.6601, ANOVA; Mean Difference (Net) = 0.021, 90% CI 2-sided [-0.059 to 0.101], Standard Error of Mean 0.048
Statistical Analysis 3: Comparison: Glimepiride 1-4 mg vs Placebo; Test type: Superiority or Other; p = 0.1412, ANOVA; Mean Difference (Net) = 0.072, 90% CI 2-sided [-0.009 to 0.152], Standard Error of Mean 0.048

4. Secondary Outcome: Number of Patients With Adverse Events
Description: Number of patients with any adverse events
Time Frame: up to 20 weeks
Population: Treated set (TS)
Measure: Number; unit: participants
Groups:
- REP - Linagliptin 5 mg: Residual effect period - Linagliptin 5 mg
- REP - Glimepiride 1-4 mg: Residual effect period - Glimepiride 1-4 mg
- Rep - Placebo: Residual effect period - Placebo
Arm/Group | Linagliptin 5 mg | Glimepiride 1-4 mg | Placebo | REP - Linagliptin 5 mg | REP - Glimepiride 1-4 mg | Rep - Placebo
Number analyzed (Participants) | 40 | 41 | 40 | 40 | 41 | 40
participants | 11 | 25 | 14 | 4 | 7 | 7

ADVERSE EVENTS:
Time Frame: 28 days treatment period + 7 days residual effect period
Description: The adverse events occurred during residual effect period (REP) were included in the frequencies.
Groups:
- Placebo: Placebo: matching Linagliptin or Glimepiride given once daily over 28 days
Arm/Group | Linagliptin 5 mg | Glimepiride 1-4 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/41 | 0/40
Other Adverse Events (participants affected / at risk) | 6/40 | 20/41 | 9/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Linagliptin 5 mg (N=40) | Glimepiride 1-4 mg (N=41) | Placebo (N=40)
Nasopharyngitis (Infections and infestations) | 1 | 6 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 16 | 1
Headache (Nervous system disorders) | 4 | 3 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.